CLINICAL TRIAL: NCT00933725
Title: Efficacy and Safety of Combined Treatment of Herbs and TCM Emotion Treatment for Women With Menopausal Syndrome: A Multiple-centered Randomized Controlled Trial
Brief Title: Efficacy and Safety of Traditional Chinese Medicine Intervention for Women With Menopausal Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2007BAI20B014; 2007BAI20B014 (Other: State Administration of TCM of China)
Record Dates: First submitted 2009-07-02; First posted 2009-07-07 (Estimated); Last update posted 2012-06-18 (Estimated); Status verified 2010-05

CONDITIONS: Menopausal Syndrome
Keywords: menopausal syndrome; TCM intervention

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TCM intervention (Experimental): Particle of compound Chinese herbs and TCM emotion treatment and tablet placebo of Tibolone
  Interventions: Other: TCM intervention
- Western intervention (Active Comparator): Tibolone and supportive psychotherapy and Particle placebo of compound Chinese herbs
  Interventions: Other: Western intervention

INTERVENTIONS:
Other: TCM intervention — Drug: Particle of compound Chinese herbs(produced by San_jiu Medical & Pharmaceutical Limited Company, Guangzhou, Guangdong Province, China), mixing with boiled water, free of decoction, taken orally, twice a day, for two months.
  One tablet placebo of Tibolone (provided by San_jiu Medical & Pharmaceutical Limited Company, Guangzhou, Guangdong Province, China, once every two days, taken orally, for two months.
  Behavioral: TCM emotion treatment: made under the guide of TCM theory, administered by qualified TCM physician, for three times in two months.
  Arms: TCM intervention
Other: Western intervention — Drug: Tibolone, (produced by Oujianong corporation, Nanjing, China), 2.5mg, once every two days, taken orally, for two months; Particle placebo of compound Chinese herbs (produced by San_jiu Medical & Pharmaceutical Limited Company, Guangzhou, Guangdong Province, China), mixing with boiled water, free of decoction, taken orally, twice a day, for two months.
  Behavioral: supportive psychotherapy, administered by qualified physician, for three times in two months.
  Arms: Western intervention

SUMMARY:
The purpose of this multiple-centered, randomized, controlled study is to investigate the efficacy and safety of a combination using herbs prescription and traditional Chinese medicine (TCM) emotion treatment in women with menopausal syndrome.

DETAILED DESCRIPTION:
Menopausal syndrome is a high incident disease which is associated with great influence in women's health and quality of life. It involves physical discomforts and emotional symptoms. Traditional Chinese medicine (TCM) theory emphasizes treating physical and emotional symptoms simultaneously viewing one person as an entirety. Herbs prescription and TCM emotion treatment is effective and safe to treat women with menopausal syndrome in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Aged 41-60;
* Amenorrhea for at least 6 months;
* Menstruation dysfunction or cessation because of age or bilateral ovariectomy;
* Hot flushes and night sweats symptoms;
* Vaginal secretion decreased with or without dyspareunia;
* Kupperman Index (KI) score ≥ 15;
* Self-rating Anxiety Scale or Self-rating Depression Scale standard score >50,but <72(standard score= scale score ×1.25);
* FSH ≥ 20 IU/L;
* Thickness of endometrium ≤0.5cm if Amenorrhea for at least 12 months;or ≤1.5cm if Amenorrhea for 6 months to 12 months;
* Meet the diagnosis criteria of TCM syndrome of liver stagnation and kidney deficiency.

Exclusion Criteria:

* With malignant tumor in reproductive system;
* With benign tumor in reproductive system and need surgery;
* Malignant tumor in mammary gland;
* Irregular vaginal bleeding for unknown reasons;
* Thickness of endometrium ≥1.5cm by ultrasound examination;
* Have used Sex hormone medicine or joined other clinical trials 3 months before;
* Allergy;
* Severe diseases (eg., of the cardiovascular, liver, kidney) or uncontrolled endocrine diseases (eg., diabetes mellitus, hyperthyreosis )
* Severe psychiatric disease diagnosed by psychiatric physician;
* Refuse informed consent.

Ages: 41 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 194 (Actual)
Dates: Start 2009-08; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Kupperman index | 2 months

SECONDARY OUTCOMES:
blood serum estradiol | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyun Wang, Bachelor, Principal Investigator — Guangzhou University of Traditional Chinese Medicine
Locations (8):
- China (8):
  - Foshan Hospital of Traditional Chinese Medicine, Foshan, Guangdong
  - Guangzhou University of Traditional Chinese Medicine, Guangzhou, Guangdong
  - Liwan Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong
  - Affiliated Hospital of Hubei College of Traditional Chinese Medicine, Wuhan, Hubei
  - Affiliated Hospital of Chengdu University of Traditional Chinese Medicine, Chengdu, Sichuan
  - Affiliated Hospital of Wenzhou Medical College, Wenzhou, Zhejiang
  - Longhua Hospital of Shanghai University of Traditional Chinese Medicine, Shanghai
  - Baokang Hospital of Tianjin University of Traditional Chinese Medicine, Tianjin